CLINICAL TRIAL: NCT00116818
Title: A Randomized, Double-blind, Parallel Group, Placebo and Active (Prednisone) Controlled, 6-week Study of the Effect of Fluticasone Furoate Aqueous Nasal Spray 100mcg QD on the Hypothalamic Pituitary Adrenocortical (HPA) Axis in Adolescents and Adults 12 to 65 Years of Age With Perennial Allergic Rhinitis (PAR)
Brief Title: A Study of GW685698X for the Treatment Of Perennial Allergic Rhinitis in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR20002
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: perennial allergic rhinitis; intranasal corticosteroid; HPA axis function; GW685698X
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X aqueous nasal spray

INTERVENTIONS:
Drug: GW685698X aqueous nasal spray

SUMMARY:
The purpose of this study is to assess the effect of an aqueous nasal spray investigational compound compared to placebo on the hypothalamic pituitary adrenocortical (HPA) axis system in adolescents and adults 12 to 65 years of age with perennial allergic rhinitis. This study can last up to 6 weeks and you will come to the clinic up to 7 times. Clinic visits include physical examinations, vital sign assessments, clinical laboratory assessments, ECGs and allergy skin testing. You will need to complete a daily diary card and spend the night in the clinic on 2 occasions to collect urine and blood samples over 24 hour periods.

DETAILED DESCRIPTION:
A randomized, double-blind, parallel group, placebo and active (prednisone) controlled, 6-week study of the effect of GW685698X aqueous nasal spray 100mcg QD on the hypothalamic pituitary adrenocortical (HPA) axis in adolescents and adults 12 to 65 years of age with perennial allergic rhinitis (PAR).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis and history of perennial allergic rhinitis.
* Must be willing to stay overnight in the clinic at the beginning and end of the study for the collection of urine and blood samples over 24 hours.
* Must comply with all study procedures and be literate.

Exclusion criteria:

* Use of tobacco products.
* Work a rotating shift.
* Significant concurrent medical conditions.
* Certain medications such as corticosteroids and allergy medications.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
HPA axis function at baseline and after 6 weeks of treatment as measured by 24 hour urine and serial serum cortisol assessments in domiciled subjects

SECONDARY OUTCOMES:
Results of adverse event, laboratory, nasal examination, vital sign, ECG and pharmacokinetic assessments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, San Antonio, Texas, United States
- GSK Investigational Site, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Patel D, Ratner P, Clements D, Wu W, Faris M, Philpot E. Lack of effect on hypothalamic-pituitary-adrenal (HPA) axis function by once-daily fluticasone furoate* nasal spray (FFNS) 110 mcg in adolescents and adults with perennial allergic rhinitis (PAR).
- [Result] Patel P, Ratner P, Clements D, Wu W, Philpot E. Twenty-four hour serum and urine cortisol data support hypothalamic-pituitary adrenocortical axis safety of once-daily fluticasone furoate*nasal spray 110mcg in adolescents and adults with perennial allerg
- [Derived] Patel D, Ratner P, Clements D, Wu W, Faris M, Philpot E. Lack of effect on adult and adolescent hypothalamic-pituitary-adrenal axis function with use of fluticasone furoate nasal spray. Ann Allergy Asthma Immunol. 2008 May;100(5):490-6. doi: 10.1016/S1081-1206(10)60476-0. PMID 18517083
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR20002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register